CLINICAL TRIAL: NCT01235260
Title: A Study of Cancer Risk Associated With Becaplermin Use in Veteran Diabetes Patients Served by the U.S. Veterans Health Administration
Brief Title: Becaplermin Use and Cancer Risk in a Patient Population of U.S. Veterans With Diabetes
Status: Completed | Type: Observational
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: Bedford Research Corporation, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: CR017497; REGRANEX-EPI-02 (Other: Johnson & Johnson Pharmaceutical Research and Development, L.L.C.)
Record Dates: First submitted 2010-11-04; First posted 2010-11-05 (Estimated); Last update posted 2016-07-19 (Estimated); Status verified 2016-07

CONDITIONS: Diabetes Mellitus; Foot Ulcer; Diabetic Foot; Diabetic Neuropathies
Keywords: REGRANEX (becaplermin); Platelet-derived growth factor BB; Cancer; Cancer incidence; Cancer mortality; Lower Extremity Diabetic Neuropathic Ulcer
MeSH Terms: conditions — Diabetes Mellitus; Foot Ulcer; Diabetic Foot; Diabetic Neuropathies; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- 001: Becaplermin users A cohort of becaplermin users (ie patients with diabetes treated with becaplermin)
  Interventions: Drug: Becaplermin users
- 002: Becaplermin nonusers A cohort of becaplermin nonusers (ie patients who are not treated with becaplermin but are similar in characteristics to patients in the becaplermin user cohort)
  Interventions: Other: Becaplermin nonusers

INTERVENTIONS:
Other: Becaplermin nonusers — A cohort of becaplermin nonusers (ie, patients who are not treated with becaplermin but are similar in characteristics to patients in the becaplermin user cohort)
  Groups: 002
Drug: Becaplermin users — A cohort of becaplermin users (ie, patients with diabetes treated with becaplermin)
  Groups: 001

SUMMARY:
The purpose of this study is to evaluate risk of cancer incidence and mortality associated with the use of REGRANEX (becaplermin) in patients with diabetes who are members of a U.S. Veterans Health Administration.

DETAILED DESCRIPTION:
This is an observational study of patients with diabetes who are eligible for care through the national Department of Veterans Affairs Health Care System (VA), representing the largest sample of older adults in an integrated health care system in the U.S. with comprehensive electronic medical records and linkable health survey data. REGRANEX (becaplermin) is topical medication used to treat lower extremity diabetic neuropathic ulcers. VA patients with diabetic foot ulcers who have no prior history of cancer who have received treatment with becaplermin will be compared to a group of similar patients who have not received treatment with becaplermin. Becaplermin users (from the time of initial dispensing of becaplermin) and becaplermin nonusers will be followed forward in time for up to 8 years to identify new cancers and cancer related deaths, with confirmation of cases through registries and medical chart review. This is an observational study; no investigational drug will be administered.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diabetic foot ulcers who are members of the U.S Department of Veterans Affairs Health Care System (VA)

Exclusion Criteria:

* History of cancer (including nonmelanoma skin cancer) prior to study entry

Max Age: 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with diabetic foot ulcers who are members of the U.S. Department of Veterans Affairs Health Care System (VA)
Sampling Method: Probability Sample
Dates: Start 2010-03; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
The number and rate of cases of incident cancers (grouped as non melanoma skin cancer, all other invasive cancers combined, and site specific cancers) in patients who have used becaplermin and patients who have not used becaplermin. | From time of recruitment beginning in October 1, 1999 until the earliest of September 30, 2007, outcome identification, or death.
The number and rate of deaths from cancer in patients who have used becaplermin and patients who have not used not used becaplermin. | From time of accrual beginning in October 1, 1999 until the earliest of September 30, 2007 or death.

SECONDARY OUTCOMES:
The number of becaplermin doses associated with risk of incident cancer and/or cancer death. | From the date of the first becaplermin dispensing beginning October 1, 1999 until the earliest of September 30, 2007, outcome identification, or death.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.